CLINICAL TRIAL: NCT05436301
Title: Turkish Validity and Reliability of Pain Catastrophizing Scale-Child (PCS-C) in Children/Adolescents With Juvenile Idiopathic Arthritis
Brief Title: Turkish Validity and Reliability of Pain Catastrophizing Scale-Child (PCS-C)
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ozge Cankaya, Principle Investigator PhD PT, Kutahya Health Sciences University
Other Study IDs: KSBU
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain; Juvenile Idiopathic Arthritis
Keywords: Chronic pain; Juvenile Idiopathic Arthritis; Pain Catastrophizing
MeSH Terms: conditions — Chronic Pain; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pain Catastrophizing Scale — Personal and disease-related inquiries of the participants will be recorded in the demographic registration form. To assess the validity of the "Pain Catastrophizing Scale-Child (PCS-C)" scale, the Pediatric Quality of Life Questionnaire (PEDSQL) 3.0 Arthritis Module, Childhood Health Assessment Questionnaire (CHAQ), and Juvenile Idiopathic Arthritis Disease Activity Score (JADAS) will be administered to the participants. In this way, the consistency of the developed scale with similar questionnaires that were previously reported to be valid will be examined. In order to determine the reliability of the "Pain Catastrophizing Scale-Child (PCS-C)" scale, test-retest will be performed at one week intervals for the participants whose treatment has not undergone any change. The consistency of the scale will be determined by the data of the participants who have the first and second scale scores. Interviews will be conducted by face-to-face method.
  Other Names: Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis Module; Childhood Health Assessment Scale (CHAQ); Juvenile Idiopathic Arthritis Disease Activity Score (JADAS)

SUMMARY:
Perception of chronic pain and related disability; occurs through the interaction of physiological and psychological processes. Pain catastrophizing is a cognitive attribution style characterized by a negative mindset and magnification of pain. Catastrophizing in children has been associated with poor functioning and higher levels of pain. Catastrophizing during the transition to adulthood is defined as an important predictor of persistent pain and central sensitivity. The number of scales assessing pain and attitudes related to pain in children is quite low. In recent years, with the adaptation of the assessment scales used for adults to children or the development of new scales, the assessment of pain and pain-related attitudes in children has begun to be provided. Pain catastrophizing scale (PCS), in 1995 Sullivan et al. for the purpose of comprehensive assessment in adults experiencing pain-related disasters. In 2003, Crombez et al. showed the validity and reliability of the scale in school-age children. For predictive validity, the scale was administered to children with chronic pain, and it was reported to predict the severity of pain and pain-related disability.

Pain Catastrophizing Scale-Child (PCS-C) scale; It is a self-report measure adapted from the Adult Pain Catastrophizing Scale used to assess negative thinking associated with pain. It contains 13 items rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true". Substances; rumination (4 items, e.g. "When [my child] has pain, I can't get him out of my mind"), magnification (3 items, e.g. the child has pain], thinking about other painful events"), and helplessness (6 items, e.g. "[My child's]] When I have pain, I feel that I cannot continue"). Items are aggregated across subscales to obtain a total score ranging from 0 to 52; higher scores are related to higher catastrophizing attitude.

The pain catastrophizing scale was originally developed in German and later validity and reliability studies were conducted in different languages. The aim of this study is to question the Turkish validity and reliability of the "Pain Catastrophizing Scale-Child (PCS-C)" scale.

DETAILED DESCRIPTION:
Now, the study is continuing. 50% of the participant were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 7-18 years old
2. Agree to participate in the study
3. Whose symptoms and medications are stable,
4. Do not have a psychiatric disease that may affect cooperation,
5. Patients with JIA who do not have heart failure and lung pathology at a level that will affect their daily living activities will be included.

Exclusion Criteria:

Participants who cannot understand and follow the instructions will be excluded from the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Juvenile Idiopathic Arthritis (JIA); It is the most common chronic rheumatic disease in childhood. It is a chronic autoimmune disease of unknown cause, in which arthritis occurs in one and/or more joints for at least 6 weeks before the age of 16. The average prevalence values found in studies conducted in various countries are between 16-150/100.000. In the study on the prevalence of JIA in our country, the rate was; It is stated as 64/100,000.
  Persistent pain is the most common and bothersome symptom of JIA, and pain in childhood arthritis is multifactorial.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Pain Catastrophizing Scale-Child (PCS-C) | 12 months
  Pain Catastrophizing Scale-Child (PCS-C); It is a self-report measure adapted from the Adult Pain Catastrophizing Scale used to assess negative thinking associated with pain. It contains 13 items rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true". Substances; rumination (4 items, e.g. "When [my child] has pain, I can't get him out of my mind"), magnification (3 items, e.g. the child has pain], thinking about other painful events"), and helplessness (6 items, e.g. "[My child's]] When I have pain, I feel that I cannot continue"). Items are aggregated across subscales to obtain a total score ranging from 0 to 52; higher scores are associated with higher catastrophizing attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Başakçı-Çalık, Prof, Study Director — Prof.
Locations (1):
- Pamukkale university, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided